CLINICAL TRIAL: NCT04327258
Title: The Influence of NPPA/NPPB Haplotype on Natriuretic Peptide Plasma Levels
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 041/09e
Record Dates: First submitted 2020-03-26; First posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Anesthesia; Surgical Procedure, Operative
Keywords: genetic association study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood (plasma and cells)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All patients: Patients undergoing elective surgery with anesthesia

SUMMARY:
Crosssectional study to analyse the genetic influence on levels of cardiac biomarkers (BNP, NT-proBNP).

DETAILED DESCRIPTION:
Background

Natriuretic peptides play an important role in risk stratification and management of patients undergoing non-cardiac surgery. However, due to genetic variability, the levels of these biomarkers may differ in individual patients with cardiac derangement. In the preoperative setting, genetic contribution to natriuretic peptide plasma level variability has not yet been determined.

Objective

The aim of this study is to assess genetic contribution to NP plasma level variability in a Swiss cohort.

Methods

Cross-sectional association study in a cohort of non-cardiac surgery patients.

This study is a Subproject of a prospective cohort study registered under the ID 041/09.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Written informed consent
* Scheduled surgery

Exclusion Criteria

* No informed consent
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2011-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Influence of NPPA/NPPB haplotype on natriuretic peptide plasma levels | Blood samples collected at start of anesthetic procedure
  Estimation of genetic effects on natriuretic peptide (BNP, NT-proBNP) plasma levels

CONTACTS AND LOCATIONS:
Overall Officials: Frank Stüber, Prof. MD, Study Chair — Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern; Ulrike M Stamer, MD, Principal Investigator — Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Inselspital, University of Bern, Bern, Switzerland